CLINICAL TRIAL: NCT02963155
Title: Prospective Study of Natural Killer Cells in Patients With Metastatic Prostate Cancer: Relationship With Survival and Response Time to Castration
Brief Title: Study of Natural Killer Cells in Patients With Metastatic Prostate Cancer: Relationship With Survival and Response Time to Castration
Acronym: NKPROSTATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NKPROSTATE-IPC 2015-019
Record Dates: First submitted 2016-11-07; First posted 2016-11-15 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Prostate Cancer
Keywords: prostate, metastatic
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metastatic prostate cancer blood samples (Experimental)
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples

SUMMARY:
Prospective research of Natural Killer cells as predictive biomarkers to stratify patients likely to have longer response time to castration.

DETAILED DESCRIPTION:
The main objective is to validate prospectively the results of a retrospective study showing a correlation between the level of NKp30 and NKp46 receptor-activators expression on the surface of NK cells and 1) the survival time, 2) the response time to castration in patients with metastatic prostate cancer.

Prospective monocenter, open-label study.

During a visit in the frame of management of the disease, a single blood sample will be collected. Patients will then have a standard care follow-up for a period of 5 years. Follow up data (death, progression) will be collected every 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with metastatic prostate cancer.
2. Aged of 18 years or more.
3. Patient in period of sensitivity to castration (patient non castrated or castration performed less than 1 year ago) and lack of progression.
4. Patient having signed an informed consent.
5. Patient affiliated to the national "Social Security" regimen or beneficiary of this regimen.

Exclusion Criteria:

1. Patient under chemotherapy treatment at the time of sampling
2. Patient under corticotherapy treatment at the time of sampling
3. Patient in emergency situation, adult subject to a measure of legal protection (placed under judicial protection, tutorship, or curatorship), or unable to give consent.
4. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study medical follow-up
5. Contraindications to study procedure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-07-07 (Actual); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Response time to castration | every 6 months during 3 years-follow up
  Time of occurrence of:
  * confirmed PSA rise + serum testosterone < 0.50 ng/mL
  * and/or radiological progression according to the modified PCWG2 criteria (progression according to the RECIST criteria v1.1 or documented by the appearance of at least 2 new lesions on the bone scan)
Survival | every 6 months during 3 and 5 years-follow up

SECONDARY OUTCOMES:
Level of alcaline phosphatase | at diagnostic (before inclusion in the study) and at time of treatment for progression in the course of 3 years-follow-up
Tumor volume | at diagnostic (before inclusion in the study)

CONTACTS AND LOCATIONS:
Overall Officials: Gwenaelle GRAVIS, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, France

REFERENCES:
- [Background] Pasero C, Gravis G, Granjeaud S, Guerin M, Thomassin-Piana J, Rocchi P, Salem N, Walz J, Moretta A, Olive D. Highly effective NK cells are associated with good prognosis in patients with metastatic prostate cancer. Oncotarget. 2015 Jun 10;6(16):14360-73. doi: 10.18632/oncotarget.3965. PMID 25961317
- [Background] Gannon PO, Poisson AO, Delvoye N, Lapointe R, Mes-Masson AM, Saad F. Characterization of the intra-prostatic immune cell infiltration in androgen-deprived prostate cancer patients. J Immunol Methods. 2009 Aug 31;348(1-2):9-17. doi: 10.1016/j.jim.2009.06.004. Epub 2009 Jun 22. PMID 19552894
- [Background] Mamessier E, Sylvain A, Thibult ML, Houvenaeghel G, Jacquemier J, Castellano R, Goncalves A, Andre P, Romagne F, Thibault G, Viens P, Birnbaum D, Bertucci F, Moretta A, Olive D. Human breast cancer cells enhance self tolerance by promoting evasion from NK cell antitumor immunity. J Clin Invest. 2011 Sep;121(9):3609-22. doi: 10.1172/JCI45816. Epub 2011 Aug 15. PMID 21841316
- See also: official website of the sponsor — http://institutpaolicalmettes.fr